CLINICAL TRIAL: NCT03857815
Title: A Phase II Study of Stereotactic Body Radiation Therapy (SBRT) Combined With Anti-PD-1 Antibody （IBI308） in Patients With Hepatocellular Carcinoma
Brief Title: Stereotactic Body Radiation Therapy Combined With Anti-PD-1 Antibody in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-HCC-SBRTPD1
Record Dates: First submitted 2019-02-24; First posted 2019-02-28 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT in combined with anti-PD-1 antibody (Experimental): HCC Patients will be received stereotactic body radiation therapy (SBRT) to primary lesions or metastatic lesions, such as liver, lung, bone, brain or lymph nodes and concurrent anti-PD-1 antibody treatment.
  Interventions: Radiation: anti-PD-1 antibody

INTERVENTIONS:
Radiation: anti-PD-1 antibody — In patients with inoperable hepatocellular carcinoma or recurrence after local or regional therapy, stereotactic body radiation therapy will be combined with anti-PD-1 antibody.
  Stereotactic body radiation therapy: SBRT is delivered to 1~5 Evaluable lesions of liver, lung, bone, brain or lymph nodes in limited fractions .
  Anti-PD-1 treatment: anti-PD-1 antibody (IBI308) is injected intravenously 200mg every three weeks.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of Stereotactic Body Radiation Therapy Combined With Anti-PD-1 Antibody in Patients in hepatocellular carcinoma.

DETAILED DESCRIPTION:
Stereotactic Body Radiation Therapy (SBRT) is an acceptable option for HCC patients not amenable to surgery or transplantation or manifested with oligometastasis. Recent studies have shown that SBRT plus immune checkpoint inhibitors may potentiate the effect of RT on tumor cell killing. The objective of this study is to evaluate the efficacy and safety of Stereotactic Body Radiation Therapy Combined With Anti-PD-1 Antibody in Patients in hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma (HCC) based on either histopathologic or cytologic findings or a diagnosis of cirrhosis and HCC with classical imaging characteristics.
* Patients including metastasis are inoperable or unresectable. Prior locoregional therapy including radiofrequency ablation, transarterial chemoembolisation, radioembolisation is allowed provided that radiologically progressive disease is demonstrated following these locoregional therapies. Lesions should be no more than five and be able to administrate SBRT, and at least one lesion is evaluable.
* The Laboratory test results must meet the following criteria:

  1. neutrophils ≥1.5×109/L
  2. Platelets ≥75×109/L
  3. Hemoglobin ≥90g/L (no blood transfusion within past 14 days)
  4. Serum Cr ≤1.5×ULN, endogenous creatinine clearance rate >60ml/min (Cockcroft-Gault formula)
  5. AST ≤2.5×ULN, ALT ≤2.5×ULN; both ALT and AST ≤5×ULN if there are liver metastasis
  6. TSH, FT3, FT4 are within ± 10% of the normal range
  7. blood coagulation functon: INR ≤2.5×ULN and APTT ≤ 1.5 ULN
* ECOG performance status: 0-1.
* Life expectancy ≥6 months.
* No history of abdominal irradiation.
* aged 18 to 75 years old are eligible.
* Patients must be able to understand and willing to sign a written informed consent document.
* Female patients within childbearing age or male patients whose sexual partners are women within childbearing age need to take effective contraceptive measures throughout the treatment period and 6 months after the treatment.

Exclusion Criteria:

* Fibrous lamina hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma.
* History of hepatic encephalopathy or liver transplantation
* Pleural effusion, ascites and pericardial effusion with clinical symptoms or needing drainage. Only a small amount of pleural effusion, ascites and pericardial effusion without symptoms could be included.
* Untreated hepatitis infection: HBV DNA>2000IU/mlor104 copy/ml, HCV RNA> 103copy/ml, both HbsAg and anti-HCV body are positive.
* Evidence with active central nervous system (CNS) metastases. Patients can be included if the CNS metastasis can be treated and the neurological symptoms can be restored to a level of ≤1 degree of CTCAE (except for residual signs or symptoms associated with CNS treatment) for at least 2 weeks before the enrollment. In addition, patients must have not be treated with a corticosteroid, or just be treated with a stable dose of ≤ 10 mg prednisone/day (or equivalent dose) or with a dose reduced to 10 mg prednisone/day;
* In the past six months, there was a history of gastrointestinal perforation and/or fistula, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive intestinal resection (partial or extensive intestinal resection with chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea.
* History of symptomatic interstitial lung disease or other conditions that may cause confusion when discovering or managing suspicious drug-related lung toxicity;
* Evidence of active pulmonary tuberculosis (TB). Patients diagnosed with active tuberculosis infection within 1 year should be excluded even if they have been treated.
* Positive test of immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
* Severe infections are in active stage or under clinical control. Severe infections occurred within 4 weeks before the first treatment, including but not limited to hospitalization due to infection, bacteremia or complications of severe pneumonia.
* Patients with active, known or suspected autoimmune diseases. Patients with the following conditions can be selected: vitiligo, type I diabetes, residual thyroid dysfunction caused by autoimmune thyroiditis that just need hormone replacement therapy, or diseases that will not relapse without external stimulating factors
* Immunosuppressive drugs have been used in the past four weeks, excluding local glucocorticoids or systemic glucocorticoids (i.e. no more than 10 mg/day prednisone or other glucocorticoids of equivalent dosage) through nasal spray, inhalation or other routes, and temporary use of glucocorticoids for the treatment of dyspnea symptoms of asthma, chronic obstructive pulmonary disease.
* Inoculation of any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.) within past 4 weeks;
* Received systemic immunostimulant therapy in the past four weeks
* Large surgical (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures have been performed in the past four weeks.
* Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary tumors may lead to higher medical risks and/or uncertainty in survival assessment.
* Some acute or chronic diseases, psychiatric disorders or abnormal laboratory test values that may lead to the result: increased risk of participating in the study or drug administration, or interfering with the interpretation of research results, and according to the judgement of the researchers, patients are classified as not eligible to participate in the study.
* Other malignant tumors were diagnosed within 5 years before the first administration, excluding cured cutaneous basal cell carcinoma, cured squamous cell carcinoma and/or cured cancer in situ. If other malignant tumors or hepatocellular carcinomas are diagnosed more than five years before administration, pathological or cytological diagnosis should be taken from recurrent and metastasis sites.
* Any prior immune checkpoint inhibition treatment with anti-PD-1/PD-L1 /PD-L2 antibody or anti-CTLA-4 antibody (or any other antibody acting on the T cell co-stimulus or checkpoint pathway)
* Patients with known sensitivity or allergy to any components of humanized anti-PD-1 antibody.
* Pregnancy and breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years to 75 Years (Adult, Older Adult)
Enrollment: 30 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression Free Survival

SECONDARY OUTCOMES:
Adverse Events | 2 years
  Adverse event (AE)、Treatment emergent adverse event(TEAE)、Serious adverse event (SAE).
OS | 2 years
  Overall survival
DCR | 2 years
  disease control rate
ORR | 2 years
  Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-Chong Zeng, PhD, Principal Investigator — Fudan University; Tian-shu Liu, PhD, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China